CLINICAL TRIAL: NCT03974230
Title: Analysis of the Genotype/Phenotype Relationship in the Fuchs' Corneal Endothelial Dystrophy in France. The French Fuchs' Follow-up Study, F3S
Brief Title: Analysis of the Genotype/Phenotype Relationship in the Fuchs' Corneal Endothelial Dystrophy in France.
Acronym: F3S
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Kyoto University, Graduate School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 18CH199; 2019-A00284-53 (Other: ANSM)
Record Dates: First submitted 2019-05-29; First posted 2019-06-04 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Fuchs Endothelial Corneal Dystrophy
Keywords: Cornea; Fuchs Endothelial Corneal Dystrophy (FECD); slit lamp; Transcription Factor 4 (TCF4); chromosome 18; genetic
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Corneal Diseases | interventions — Blood Specimen Collection; Slit Lamp

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample will be performed (genetic analyses).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Fuchs Endothelial Corneal Dystrophy (FECD): Patients with Fuchs Endothelial Corneal Dystrophy (FECD). They will have a collection of datas and a blood sample.
  Interventions: Other: Collection of datas; Biological: blood sample
- Control group: Witness will be included in control group. They will have a blood sample and slit lamp examination.
  Interventions: Biological: blood sample; Other: slit lamp examination

INTERVENTIONS:
Other: Collection of datas — Collection of datas of examination for diagnosis and follow-up of the Fuchs Endothelial Corneal Dystrophy (FECD) including slit lamp results will be performed.
  Groups: Patients with Fuchs Endothelial Corneal Dystrophy (FECD)
Biological: blood sample — Blood sample will be performed (genetic analyses).
Other: slit lamp examination — Slit lamp examination will be performed.
  Groups: Control group

SUMMARY:
The pathophysiology of the most common corneal endothelial dystrophies (Fuchs' Corneal Endothelial Dystrophy (FECD)) is beginning to be dismembered. One of the most common genetic anomalies is a triplet repetition in one of the introns of the Transcription Factor 4 (TCF4) gene located on chromosome 18. However, the number of repetitions varies greatly from one patient to another.

DETAILED DESCRIPTION:
The intent of that study was to analyse if there is a relationship between the number of triplet repetitions and the rate of disease progression. This knowledge would make it possible to personalize the care.

ELIGIBILITY:
Inclusion Criteria:

For patient group:

* >18 years old
* affiliated with or entitled to a social security scheme
* having received informed information about the study and having co-signed, with the investigator, a consent to participate in the study
* with an Fuchs Endothelial Corneal Dystrophy (FECD) certified by slit lamp examination

For control group:

* >18 years old
* affiliated with or entitled to a social security scheme
* having received informed information about the study and having co-signed, with the investigator, a consent to participate in the study

Exclusion Criteria:

For patient group:

* Patients under guardianship or curatorship
* Patient planning to move within the year
* With no evidence of ophthalmological pathology requiring intraocular surgery within one year of the first visit
* Better initial corrected visual acuity <1/10
* Not having had intraocular surgery in the 6 months prior to inclusion (after 6 months, the endothelium is considered stabilized)
* Not having any other progressive pathology responsible for a decrease in visual acuity (significant cataract Lens Opacities Classification System (LOCS) >2 ; progressive retinal pathology, in particular age-related macular degeneration, unstabilized macular edema)

For control group:

* Patients under guardianship or curatorship
* with an Fuchs Endothelial Corneal Dystrophy (FECD) certified by slit lamp examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There are 2 cohorts: patient and control.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Visual acuity | Year: 0 and 1
  Correlation between visual acuity measured before noon eye by eye of ETDRS scale (international standardized Early Treatment Diabetic Retinopathy Study scale) results and number of CTG triplet repetitions in the intron of the Transcription Factor 4 (TCF4) gene.

SECONDARY OUTCOMES:
CTG triplet repetitions in the intron of the Transcription Factor 4 (TCF4) gene | Year: 0 and 1
  Analysis number of CTG triplet repetitions in the intron of the Transcription Factor 4 (TCF4) gene.
Mutation rs613872 | Year: 0 and 1
  Analysis frequency of the mutation rs613872 in the intron of the Transcription Factor 4 (TCF4) gene.
Other mutation | Year: 0 and 1
  Analysis frequency of the other mutation type nucleotide polymorphisms in the intron of the Transcription Factor 4 (TCF4) gene.
Refraction with the auto-refractor tonometry | Year: 0 and 1
  Analysis refraction with the auto-refractor tonometry non-contact air.
ETDRS scale (Early Treatment Diabetic Retinopathy Study scale) in a controlled glare situation | Year: 0 and 1
  Correlation between visual acuity measured before noon eye by eye on the ETDRS scale (Early Treatment Diabetic Retinopathy Study scale) in a controlled glare situation.
  ETDRS (Early Treatment Diabetic Retinopathy Study) scale will be allowed to measure visual acuity uses an eye chart with 5 letters per line. The scores range from 0 (no letters read correctly) to 100 (all letters read correctly).
interferometry, tear meniscus height, Non Invasive Break-Up Time (NIBUT) and meibography | Year: 0 and 1
  Correlation between interferometry, tear meniscus height, Non Invasive Break-Up Time (NIBUT) and meibography results.
Corneal thickness in Optical Coherence Tomography (OCT) | Year: 0 and 1
  Comparison corneal thickness in Optical Coherence Tomography (OCT).
Reflectivity results measure by Optical Coherence Tomography (OCT) | Year: 0 and 1
  Comparison reflectivity results measure by Optical Coherence Tomography (OCT). Optical Coherence Tomography (OCT) is an imaging technique, which is able to produce, in vivo, cross-sectional images of lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles THURET, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dorado Cortez O, Fleischmann Caruso D, Crouzet E, Poinard S, Trone MC, Gain P, Okumura N, Koizumi N, Thuret G. Assessing Corneal Tomographic Changes in Fuchs Endothelial Corneal Dystrophy Over 1 Year: Scheimpflug Versus Anterior Segment Optical Coherence Tomography. Cornea. 2024 Dec 11;44(9):1127-1135. doi: 10.1097/ICO.0000000000003771. PMID 39661178
- [Derived] Dorado-Cortez O, Crouzet E, Trone MC, Gain P, He Z, Vaitinadapoule H, Mentek M, Mascarelli F, Poinard S, Yasunaga M, Nishiuchi G, Koizumi N, Okumura N, Thuret G. Change in Visual Acuity of Patients With Fuchs Endothelial Corneal Dystrophy Over 1 Year. Cornea. 2024 Oct 1;43(10):1207-1215. doi: 10.1097/ICO.0000000000003590. Epub 2024 Jul 9. PMID 39288343